CLINICAL TRIAL: NCT00220922
Title: An Open-Label, Randomized, Single Cross-Over Study of Isopropyl Alcohol Wipes Versus No Injection Site Preparation on Local Injection Site Reactions Among Persons With Multiple Sclerosis Who Perform Daily Injections of Copaxone®
Brief Title: A Study to Evaluate the Impact on Skin (Injection Site) Reactions of Using Alcohol Wipes Prior to Daily Injections of Copaxone®.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Neuroscience, Inc. (Industry)
Responsible Party: Thomas Smith, M.D., Vice President, Medical Affairs, Teva Neuroscience
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PM013
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Multiple Sclerosis
Keywords: Copaxone
MeSH Terms: conditions — Multiple Sclerosis | interventions — Ethanol; Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): injection site reactions with the use of alcohol wipes prior to performing the patients' daily Copaxone® injection
  Interventions: Procedure: Alcohol Wipes vs. No Alcohol Wipes
- 2 (Experimental): injection site reactions without the use of alcohol wipes prior to performing the patients' daily Copaxone® injection
  Interventions: Procedure: Alcohol Wipes vs. No Alcohol Wipes

INTERVENTIONS:
Procedure: Alcohol Wipes vs. No Alcohol Wipes
  Other Names: Copaxone

SUMMARY:
This study is designed to compare injection site reactions with or without the use of alcohol wipes prior to performing the patients' daily Copaxone® injection.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 18 years of age or older
* Diagnosis of RRMS
* Beginning or recently (within 3 months) began self-injecting Copaxone® subcutaneously

Exclusion Criteria:

* Unable to perform subcutaneous self-injection
* Pregnant, or trying to become pregnant, or breast feeding during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-08; Primary Completion 2005-10 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Total number of local injection site reactions (LISRs) noted at 5-minutes post-injection | four weeks of Period 1 and the four weeks of Period 2

SECONDARY OUTCOMES:
The total number of LISRs noted at 2-minutes post-injection The total number of LISRs noted immediately after injection | four weeks of Period 1 and the four weeks of Period 2

CONTACTS AND LOCATIONS:
Overall Officials: MerriKay Oleen-Burkey, Ph.D., Study Director — Teva Neuroscience, Inc.